CLINICAL TRIAL: NCT06787443
Title: A Randomized, Placebo Controlled Clinical Study to Examine the Clinical Benefits of an Oral Product in Subjects With Menopausal Symptoms Including Vasomotor Symptoms
Brief Title: Randomized Placebo Controlled Clinical Study of an Oral Product in Subjects With Menopausal Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olly, PBC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: UNLV20240222
Record Dates: First submitted 2024-11-21; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Menopausal Symptoms
MeSH Terms: interventions — Dietary Supplements; gamma-Aminobutyric Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Dietary Supplement with Actives (Active Comparator)
  Interventions: Dietary Supplement: Dietary Supplement with Proprietary Herbal Extract Blend and GABA

INTERVENTIONS:
Dietary Supplement: Placebo — Eligible subjects will receive Placebo to take daily for five weeks
  Arms: Placebo
Dietary Supplement: Dietary Supplement with Proprietary Herbal Extract Blend and GABA — Eligible subjects will receive active product to take daily for five weeks
  Arms: Dietary Supplement with Actives

SUMMARY:
The objective of this study is to assess the safety and effectiveness of a dietary supplement for symptom relief in subjects with menopausal symptoms over the course of five weeks of continuous daily use.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Females aged 40 to 65 years,
* Self-reporting menopausal symptoms (> 5 hot flushes per day) and have been present for a minimum of previous 60 days prior to baseline visit.
* Reporting a variable cycle length of > 7 days different from normal
* BMI 20-40 kg/m2
* Able to read, understand, and complete the study questionnaire and records.
* Able to understand the study procedures.
* Able to comply with all study requirements.
* Written informed consent to participate in the study.
* Willingness to actively participate in the study and to come to the scheduled visits.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Immune insufficiency
* Women of childbearing potential including those still having a menstrual cycle on a regular basis who are not perimenopausal, menopausal or post-menopausal.
* History of hysterectomy
* Women on hormone replacement therapy
* Use of systemic corticosteroids or immunosuppressant drugs.
* Other diseases or medications that might directly interfere in the study or put the subject's health under risk.
* Employees of the institute
* Cardiovascular-, chronic liver-, thyroid or kidney diseases; a history of cancer; a disease or condition that could influence the participants' ability to follow the study protocol,
* Alcohol or drug abuse,
* Use of hormonal contraceptives within the last 3 months
* BP ≥160/110 mmHg
* Oophorectomy or amenorrhea > two years

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2024-05-10 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Changes of symptom scores in Daily Dairy | from enrollment to the end of study at five weeks
  To assess changes in symptom scores attained from product use in subjects with menopausal symptoms, including acute effects
Changes of symptom scores in Mobile Application | from enrollment to the end of study at five weeks
  To assess changes in symptom scores attained from product use in subjects with menopausal symptoms, including acute effects

SECONDARY OUTCOMES:
Changes in Menopause-Specific Quality of Life (MENQOL) Scores | from enrollment to the end of study at five weeks
  To assess changes in mood and quality of life scores of the product compared to placebo
Changes in Green Climacteric Scale (GCS) Scores | from enrollment to the end of study at five weeks
  To assess changes in mood scores of the product compared to placebo
Changes in Perceived Stress Scale (PSS) Scores | from enrollment to the end of study at five weeks
  To assess changes in mood scores of the product compared to placebo
Changes in Profile of Mood States (POMS) Scores | from enrollment to the end of study at five weeks
  To assess changes in mood scores of the product compared to placebo
Changes in Pittsburgh Sleep Quality Index (PSQI) Scores | from enrollment to the end of study at five weeks
  To assess changes in sleep scores of the product compared to placebo

CONTACTS AND LOCATIONS:
Locations (1):
- See Final Report, San Francisco, California, United States